CLINICAL TRIAL: NCT02790996
Title: Multi-centre, Randomised, Open Label, Phase IIb Study to Compare the Efficacy, Safety and Pharmacokinetics (PK) of an Optimised Dosing to a Standard Dosing Regimen of Vancomycin in Neonates and Infants Aged ≤ 90 Days With Late Onset Bacterial Sepsis Known or Suspected to be Caused by Gram-positive Microorganisms
Brief Title: Neonatal Vancomycin Trial
Acronym: NeoVanc
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Planned interim analysis yielded different event rate affecting sample size and ability to recruit sufficient numbers within remaining trial time frame
Sponsor: PENTA Foundation (Network)
Collaborators: St George's, University of London (Other); Hopital Universitaire Robert-Debre (Other); University of Tartu (Other); Consorzio per Valutazioni Biologiche e Farmacologiche (Other); University of Liverpool (Other); Therakind limited (Unknown); Bambino Gesù Hospital and Research Institute (Other); Servicio Madrileño de Salud, Madrid, Spain (Other); Aristotle University Of Thessaloniki (Other); Cardiff University (Other); SYNAPSE Research Management Partners S.L (Unknown); European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeoVanc
Record Dates: First submitted 2016-04-07; First posted 2016-06-06 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Late Onset Neonatal Sepsis
Keywords: sepsis; neonate; vancomycin
MeSH Terms: conditions — Neonatal Sepsis; Sepsis | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vancomycin - Optimised Regimen (Experimental): A single loading dose of 25 mg/kg followed by a maintenance dose of:
  Postmenstrual age ≤ 35 weeks - 15 mg/kg 12 hourly; Postmenstrual age > 35 weeks - 15 mg/kg 8 hourly
  Interventions: Drug: Vancomycin
- Vancomycin - Standard Regimen (Active Comparator): Postmenstrual age < 29 weeks - 15 mg/kg given 24 hourly; Postmenstrual age 29 - 35 weeks - 15 mg/kg 12 hourly; Postmenstrual age > 35 weeks - 15 mg/kg 8 hourly
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Vancomycin is an antibiotic used to treat a number of bacterial infections.It is recommended intravenously as a treatment for complicated skin infections, bloodstream infections, endocarditis, bone and joint infections, and meningitis caused by methicillin-resistant S. aureus.

SUMMARY:
The study aims to compare the efficacy, safety and pharmacokinetics (PK) of an optimised dosing to a standard dosing regimen of vancomycin in neonates and infants aged ≤ 90 days with late onset bacterial sepsis known or suspected to be caused by Gram-positive microorganisms

DETAILED DESCRIPTION:
Detailed objectives of the study are:

* To compare the efficacy of an optimised vancomycin dosing regimen to a standard vancomycin dosing regimen in patients with late onset, bacterial sepsis, known or suspected to be caused by Gram-positive microorganisms.
* To compare the safety of vancomycin (including renal and hearing safety) by allocation group in the intention to treat (ITT) population
* To describe the PK parameters according to vancomycin dosing regimen and outcome using population PK modelling in the ITT population
* To describe PK/PD in terms of the probability of target attainment (PTA) with different vancomycin dosing regimens in the ITT and per protocol (PP) populations
* To describe outcomes and duration of therapy at the end of vancomycin treatment and at the short term follow-up visit by allocation group in the ITT and PP populations
* To compare the clinical outcome to the antibacterial susceptibility of infecting organisms
* To compare colonisation by resistant microorganisms (e.g. vancomycin-resistant enterococci (VRE)) and Candida spp. by allocation group at baseline, TOC and short-term follow-up
* To validate across multiple centres a host biomarker panel to allow improved diagnosis of bacterial sepsis and monitor response to antibacterial therapy

ELIGIBILITY:
Inclusion Criteria:

* Postnatal age ≤ 90 days AND
* Postnatal age ≥ 72 hours at onset of sepsis AND
* Clinical sepsis as defined by presence of any three clinical or laboratory criteria from the list below OR
* Confirmed, significant bacterial sepsis as defined by positive culture with a Gram-positive bacterium from a normally sterile site and at least one clinical or one laboratory criterion from the list below, in the 24 hours before randomisation

Clinical criteria

* hyper- or hypothermia,
* hypotension or impaired peripheral perfusion or mottled skin,
* apnoea or increased oxygen requirement or increased requirement for ventilatory support,
* bradycardic episodes or tachycardia,
* worsening feeding intolerance or abdominal distension,
* lethargy or hypotonia or irritability

Laboratory criteria:

* white blood cell (WBC) count < 4 or > 20 x 109 cells/L
* immature to total neutrophil ratio (I/T) > 0.2
* platelet count < 100 x 109/L
* C-reactive protein (CRP) > 10 mg/L
* glucose intolerance as defined by a blood glucose value > 180 mg/dL (> 10 mmol/L) when receiving normal glucose amounts (8 - 15 g/kg/day)
* metabolic acidosis as defined by a base excess (BE) < -10 mmol/L (-10 mEq/L) or a blood lactate value > 2 mmol/L

Exclusion Criteria:

* Administration of any systemic antibiotic regimen for more than 24 hours prior to randomisation, unless the change is driven by the apparent lack of efficacy of the original regimen
* Treatment with vancomycin for ≥ 24 hours at any time within 7 days of enrolment
* Known toxicity, hypersensitivity or intolerance to vancomycin
* Known renal impairment with urinary output < 0.7 ml/kg/hour for 24 hours or a creatinine value ≥ 100 µmol/L (1.13 mg/dL)
* Patient receiving (or planned to receive) haemofiltration, haemodialysis, peritoneal dialysis, extracorporeal membrane oxygenation (ECMO) or cardiopulmonary bypass
* Severe congenital malformations where the infant is not expected to survive for more than 3 months
* Patient known to have S. aureus (MSSA or MRSA) bacteraemia
* Patient with osteomyelitis, septic arthritis, urinary tract infection (UTI) or meningitis
* Patient with high suspicion of/confirmed sepsis caused by Gram-negative organisms or fungi
* Other situations where the treating physician considers a different empiric antibiotic regimen necessary
* Current participation in any other clinical study of an investigational medicinal product (IMP)

Post-randomisation exclusions

• Any participant found to have Gram-negative or fungal sepsis, osteomyelitis, septic arthritis, UTI, meningitis or S. aureus (MSSA or MRSA) bacteraemia after randomisation will be excluded from analysis. Participants who have received at least one dose of study vancomycin will be followed up for safety

Ages: 72 Hours to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 242 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Successful outcome at Test of Cure visit | 10±1 days after End of Actual Vancomycin Therapy
  Patient is alive AND has a successful outcome at the end of actual vancomycin therapy AND the patient has not had a clinically or microbiologically significant relapse or new infection.

SECONDARY OUTCOMES:
Clinically or microbiologically significant relapse or new infection requiring treatment with any other antibiotic for more than 24 hours | 10±1 days after the End of Actual Vancomycin Treatment
Successful outcome at Visit 4 or End of Actual Vancomycin Therapy including total duration of vancomycin therapy | Day 5±1 or Day 10±2
Abnormal renal function tests at the Short-term Follow-Up Visit | 30±5 days post-initiation of vancomycin therapy
Abnormal hearing screening test | By Day 90 post-initiation of vancomycin therapy
Comparative safety of vancomycin (relating to the number of treatment-related adverse events other than those associated with renal function and hearing) at Short Term Follow-Up Visit | 30±5 days post-initiation of vancomycin therapy
Pharmacokinetic parameters of vancomycin using population PK modelling by allocation group | Up to 2 years (final data collection date for outcome measure)
  Area under the plasma concentration time curve - AUC (mg*hour/L)
Probability of target attainment (PTA) with different study regimens | Up to 2 years (final data collection date for outcome measure)
  Different bacteriological targets will be tested, based on the MIC of different bacteria of interest with level of sensitivity. Simulations based on the vancomycin popPK model will be conducted to define the number of patients in the different allocation groups reaching the predefined targets when modifying the dose.
Relationship between CoNS species and duration of treatment and CRP response | Day 5±1 or Day 10±1
Gut colonisation by vancomycin resistant organisms at baseline, Test of Cure Visit and Short-term Follow-Up Visit | Baseline, 10±1 days after end of vancomycin therapy, 30±5 days post-initiation of vancomycin therapy
Skin colonisation and resistance patterns before and after vancomycin treatment | Baseline, 10±1 days after end of vancomycin therapy, 30±5 days post-initiation of vancomycin therapy
Assessment of changes in host biomarker panel profiles from baseline to End of Actual Vancomycin Therapy and the relationship between host biomarker and duration of treatment | Day 3 and Day 5±1, Day 10±1 (standard arm only)
  Functional molecular units based on a multimarker panel - a set of 52 biomarkers will be performed as a classifier with high accuracy and specificity in predicting bacterial infection

CONTACTS AND LOCATIONS:
Overall Officials: Mike Sharland, MD, FRCPCH, Study Chair — St George's, University of London
Locations (18):
- Estonia (2):
  - Tallinn's Children's Hospital, Tallinn
  - Paediatric Intensive Care Unit, Clinicum of the University of Tartu, Tartu
- Greece (7):
  - Aghia Sophia Children's Hospital (A), Athens
  - Aghia Sophia Children's Hospital (B), Athens
  - Aghia Sophia Children's Hospital (C), Athens
  - Kyriakou Children's Hospital, Athens
  - General University Hospital Attikon, Chaïdári
  - Hippokration Hospital - Department of Neonatology, Thessaloniki
  - Papageorgiou 2nd Department of Neonatology, Thessaloniki
- Italy (5):
  - Ospedale "Di Venere" - Carbonara di Bari, Bari
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Policlinico San Matteo, Pavia
  - Ospedale Pediatrico Bambino Gesu', Rome
- Spain (3):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital Materno Infantil, La Paz, Madrid
- St Mary's Hospital, Manchester, United Kingdom

REFERENCES:
- [Background] Hill LF, Turner MA, Lutsar I, Heath PT, Hardy P, Linsell L, Jacqz-Aigrain E, Roilides E, Sharland M; NeoVanc Consortium. An optimised dosing regimen versus a standard dosing regimen of vancomycin for the treatment of late onset sepsis due to Gram-positive microorganisms in neonates and infants aged less than 90 days (NeoVanc): study protocol for a randomised controlled trial. Trials. 2020 Apr 15;21(1):329. doi: 10.1186/s13063-020-4184-8. PMID 32293527
- [Derived] Hill LF, Clements MN, Turner MA, Dona D, Lutsar I, Jacqz-Aigrain E, Heath PT, Roilides E, Rawcliffe L, Alonso-Diaz C, Baraldi E, Dotta A, Ilmoja ML, Mahaveer A, Metsvaht T, Mitsiakos G, Papaevangelou V, Sarafidis K, Walker AS, Sharland M; NeoVanc Consortium. Optimised versus standard dosing of vancomycin in infants with Gram-positive sepsis (NeoVanc): a multicentre, randomised, open-label, phase 2b, non-inferiority trial. Lancet Child Adolesc Health. 2022 Jan;6(1):49-59. doi: 10.1016/S2352-4642(21)00305-9. Epub 2021 Nov 26. PMID 34843669